CLINICAL TRIAL: NCT00472043
Title: A Multicentre, Phase III, Double Blind Study of Photodynamic Therapy (PDT) With Metvix® 160 mg/g Cream in Comparison to PDT With Placebo Cream in Participants With Primary Nodular Basal Cell Carcinoma
Brief Title: PDT With Metvix 160 mg/g Cream Versus PDT With Placebo Cream in Participants With Primary Nodular Basal Call Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC T308/00
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-02

CONDITIONS: Basal Cell Carcinoma
Keywords: Nodular Basal Cell Carcinoma; Basal Cell Carcinoma; Photodynamic therapy (PDT); Metvix; Histological verification; PDT with Metvix cream; PDT with Placebo cream
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — 1-phenyl-3,3-dimethyltriazene; methyl 5-aminolevulinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metvix® cream 160 milligram per gram (Experimental): Methyl aminolevulinate hydrochloride 160 milligram (mg)/gram (g) cream were received by participants with primary nodular basal cell carcinoma. A thick layer of study cream was applied directly on the lesion and on 5 mm of the surrounding tissue. An approximately 1 mm thick layer of cream was applied to cover the lesion completely. The study cream was applied for at least 3 hours followed by illumination using non-coherent red (570-670 nm) light at a fluence of 50- 75 J/cm^2.
  Interventions: Drug: PDT with Metvix 160 mg/g cream
- Placebo (Placebo Comparator): Participants with primary nodular basal cell carcinoma received Metvix® matching placebo cream. A thick layer of study cream was applied directly on the lesion and on 5 mm of the surrounding tissue. An approximately 1 mm thick layer of cream was applied to cover the lesion completely. The study cream was applied for at least 3 hours followed by illumination using non-coherent red (570-670 nm) light at a fluence of 50- 75 J/cm^2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PDT with Metvix 160 mg/g cream
  Arms: Metvix® cream 160 milligram per gram
Drug: Placebo
  Arms: Placebo

SUMMARY:
Photodynamic therapy (PDT) was the selective destruction of abnormal cells through light activation of a photosensitiser in the presence of oxygen. These cells accumulated more photosensitiser than normal cells. The photosensitiser generated reactive oxygen species upon illumination.

For skin diseases, there had been an increasing interest in using precursors of the endogenous photosensitiser protoporphyrin IX (PpIX). The most commonly used precursors had been 5-aminolevulinic acid (ALA) and its derivatives. The present test drug, Metvix®, contained the methyl ester of ALA, which penetrated the lesions well and shows high lesion selectivity .

In vitro studies of animal and human tissues had shown significant intracellular formation of photoactive porphyrins after addition of Metvix®. The increased levels of photoactive porphyrins induced cytotoxic effects in tumour cells after photoactivation.

The primary objective was to compare PDT with Metvix® cream to PDT with placebo cream in terms of participant complete response rates based on histologically verified disappearance of the lesions at 6 months after last treatment cycle.

Secondary objectives were to compare the two treatments in terms of histological and clinical mean participant response weighted by the number of lesions within a participant, lesion response rates across participants, clinical complete participant response, cosmetic outcome and adverse events.

DETAILED DESCRIPTION:
A participant was randomised to PDT with Metvix® cream or PDT with placebo cream. All eligible Basal cell carcinoma (BCC) lesions within a participant had got the same treatment. All participants got two consecutive treatments one week apart. At the 3-months follow-up visit, lesions with no clinical response or progression had been surgically excised. Lesions with partial response (50% or greater reduction on lesion area) had been re-treated, if they do not show complete response three months later they would have been be surgically excised. Lesions with complete response had been surgically excised 6 months after the first or second PDT cycle. All excised tissue specimens had been histologically examined.

ELIGIBILITY:
Inclusion Criteria:

A participant with primary, nodular BCC lesion(s) suitable for entry is defined as a participant with

* Clinically diagnosed primary nodular BCC lesion(s).
* Histologically confirmed diagnosis of BCC.
* BCC lesions suitable for simple excision surgery.
* Males or females above 18 years of age.
* Written informed consent.

Exclusion Criteria:

A participant that is ineligible for inclusion is a participant fulfilling any of the following criteria:

* Participants with porphyria.
* Participant with Gorlin's syndrome.
* Participant with Xeroderma pigmentosum.
* Participants concurrently receiving immunosuppressive medication.
* Participants with a history of arsenic exposure.
* Known allergy to Metvix®, a similar PDT compound or excipients of the cream.
* Participation in other clinical studies either concurrently or within the last 30 days.
* Pregnant or breast-feeding: All women of child-bearing potential must use adequate contraception (e.g. barrier methods, oral contraceptives or intrauterine device) during the treatment period and one month thereafter. In addition, they must have a negative pregnancy test prior to treatment.
* Conditions associated with a risk of poor protocol compliance.

Lesion Exclusion Criteria:

* A nodular BCC lesion in periorbital area, ears and nasolabial fold.
* A nodular BCC lesion with the longest diameter less than 6 mm or larger than 15 mm in face/scalp, larger than 20 mm on extremities and neck and larger than 30 mm on truncus.
* Pigmented nodular BCC lesion(s).
* Morpheaform nodular BCC lesion(s).
* Infiltrating nodular BCC lesion(s).
* Prior treatment of the BCC lesion(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2000-10-01 (Actual); Primary Completion 2002-09-30 (Actual); Study Completion 2002-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Foley, MD, Principal Investigator — Department of Dermatology, St. Vincent's Hospital Melbourne
Locations (7):
- Australia (7):
  - Dept. of Dermatology, Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Dermatology Dept., St. George Hospital, Kogarah, New South Wales
  - Dermatology Centre, Liverpool, New South Wales
  - Dr. Michael Freeman, Benowa, Queensland
  - Dermatology Dept., Princess Alexandra Hospital, Woolloongabba, Queensland
  - Department of Dermatology, St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in Australia between 1 October 2000 to 30 September 2002.
Pre-assignment Details: A total of 66 participants were included in this study.
Period: Overall Study
Arm/Group | Metvix® Cream 160 Milligram Per Gram | Placebo
Started | 33 | 33
Completed | 31 | 33
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention to Treat (ITT) population that included all treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metvix® Cream 160 Milligram Per Gram | Placebo | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (10) | 66 (11) | 68 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 22 | 27 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 33 | 33 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Histologically Confirmed Complete Response (CR)
Description: Complete Response (CR) was defined as 100 percentage of the lesions within the participant having negative findings for nodular basal cell carcinoma (BCC) in the histological examination. Histological examination included evaluation of all the microscopical slides from the excised tissue for presence of malignant basal cells. Complete response was defined as complete disappearance of lesion. Percentage of participants with histologically confirmed complete response were reported.
Time Frame: up to 6 months
Population: Intent to treat (ITT) population that included all treated participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Metvix® Cream 160 Milligram Per Gram | Placebo
Number analyzed (Participants) | 33 | 33
percentage of participants | 67 [48 to 82] | 18 [7 to 36]
Statistical Analysis 1: Comparison: Metvix® Cream 160 Milligram Per Gram vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level

2. Secondary Outcome: Percentage of Lesions Per Participant: Histologically Confirmed Participant Weighted Response
Description: Histological response weight means no signs of malignant basal cells in all microscopical slides containing excised tissue. The histologically confirmed participant weighted response, weighted by percentage of lesions per participant are reported in this outcome measure. Number of lesions per participant with-in treatment group were calculated in following way: ni = number of lesions within 1 participant, ci= number of lesions in complete response within 1 participant, xi= 100%. ci/ni= response rate within one participant, Nt= number of participant within one treatment, nt=number of lesions with-in one treatment, wi=ni/nt= weight for one participant with Nt Σ wi (i=1) = 1 for each treatment.
Time Frame: Up to 3 months
Population: ITT Population that included all treated participants
Measure: Mean (Standard Deviation); unit: Percentage of lesions per participant
Units Other Than Participants: Lesions
Arm/Group | Metvix® Cream 160 Milligram Per Gram | Placebo
Number analyzed (Participants) | 33 | 33
Number analyzed (Lesions) | 34 | 36
Percentage of lesions per participant | 67.6 (8.3) | 19.4 (6.7)

3. Secondary Outcome: Histological Lesion Response
Description: Histological examination included from the excised tissue were examined for presence of malignant basal cells, where complete response (CR) was no signs of malignant basal cells and non-CR was evidence of malignant basal cells
Time Frame: Up to 3 months
Population: ITT population included all treated participants
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Metvix® Cream 160 Milligram Per Gram | Placebo
Number analyzed (Participants) | 33 | 33
Number analyzed (Lesions) | 34 | 36
Lesions
  Lesions in CR | 23 | 7
  Lesions in non-CR | 8 | 29
  Missing | 3 | 0

4. Secondary Outcome: Percentage of Participants With Clinically Confirmed Participant Complete Response (CR)
Description: A CR to treatment was documented clinically by visual evaluation and palpation. The on-site investigator evaluated the lesion response by comparing with the lesion size before treatment using the following definitions: CR - complete disappearance of a lesion. Partial response (PR) -the longest diameter of the lesion is reduced by 50% or more. No response (NR) - the longest diameter of the lesion is less than 50% reduced. Progression - the longest diameter is increased by 20% or more.
Time Frame: Up to 9 months
Population: ITT population that includes all treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Metvix® Cream 160 Milligram Per Gram | Placebo
Number analyzed (Participants) | 33 | 33
percentage of participants | 82 | 24

5. Secondary Outcome: Cosmetic Outcomes for Lesions Assessed by Investigator
Description: Cosmetic outcome for those lesions with complete histological response was assessed by both the investigator and by the participant. Cosmetic outcome was assessed with regards to occurrence of the following signs or symptoms like scarring, atrophy, induration, redness, and change in pigmentation. The cosmetic outcome was graded as excellent: no scarring, atrophy or induration, and no or slight occurrence of redness or change in pigmentation compared to adjacent skin; good: no scarring, atrophy or induration but moderate redness or change in pigmentation compared to adjacent skin; fair: slight to moderate occurrence of scarring, atrophy or induration; poor: extensive occurrence of scarring, atrophy or induration.
Time Frame: Up to 3 months
Population: ITT population that includes all treated participants
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Metvix® Cream 160 Milligram Per Gram | Placebo
Number analyzed (Participants) | 33 | 33
Number analyzed (Lesions) | 23 | 7
Lesions
  Investigator: Excellent | 13 | 2
  Investigator: Good | 8 | 3
  Investigator: Fair | 1 | 1
  Investigator: Not Applicable | 1 | 1

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and AEs Leading to Discontinuation
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily had a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A SAE was any untoward medical occurrence that at any dose: results in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect.
Time Frame: Up to 6 months
Population: The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix® Cream 160 Milligram Per Gram | Placebo
Number analyzed (Participants) | 33 | 33
Participants
  Serious adverse events | 1 | 2
  Adverse events leading to discontinuation | 1 | 0

7. Secondary Outcome: Cosmetic Outcomes for Lesions Assessed by Participants
Description: as for outcome 5
Time Frame: Up to 3 months
Population: ITT population that includes all treated participants
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Metvix® Cream 160 Milligram Per Gram | Placebo
Number analyzed (Participants) | 33 | 33
Number analyzed (Lesions) | 23 | 7
Lesions
  Participants: Excellent | 14 | 5
  Participants: Good | 8 | 1
  Participants: Fair | 0 | 0
  Participants: Not Applicable | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Analysis was performed on safety population: randomized participants who applied the study medication at least once.
Arm/Group | Metvix® Cream 160 Milligram Per Gram | Placebo
All-Cause Mortality (participants affected / at risk) | 1/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/33 | 2/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metvix® Cream 160 Milligram Per Gram (N=33) | Placebo (N=33)
Carcinoma Bile Duct (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes